CLINICAL TRIAL: NCT04917965
Title: Thromboelastographic Profile in Healthy Newborns and Infants of Diabetic Mothers Using TEG6s
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 262407
Record Dates: First submitted 2021-06-02; First posted 2021-06-08 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Thromboelastography; Coagulation; Fetus or Newborn; Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1; Diabetes, Gestational
Keywords: thromboelastography; infant of diabetic mother; coagulation profile
MeSH Terms: conditions — Thrombosis; Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1; Diabetes, Gestational

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Term Neonates: Infants born at 37 weeks gestational age or greater born to mothers of any age with uncomplicated pregnancies. Following delivery, cord blood obtained from the placental portion of the umbilical cord will be used for analysis. To assure appropriate dilution, a hematocrit will be measured at the time of blood collection using a blood gas machine for prompt results. Sample blood will immediately be taken by the investigators from the delivery hospital to the children's hospital where the following clotting studies will be performed: PT, aPTT, fibrinogen, platelet count, platelet mapping, and TEG6s. Specimens will be transported utilizing Specimen Transport Guidelines.
  Interventions: Other: Laboratory clotting studies
- Term infants of diabetic mothers: Infants born at 37 weeks gestational age or greater to mothers of any age with gestational diabetes or Type 1 or Type 2 diabetes, managed with either diet or insulin. Following delivery, cord blood obtained from the placental portion of the umbilical cord will be used for analysis. To assure appropriate dilution, a hematocrit will be measured at the time of blood collection using a blood gas machine for prompt results. Sample blood will immediately be taken by the investigators from the delivery hospital to the children's hospital where the following clotting studies will be performed: PT, aPTT, fibrinogen, platelet count, platelet mapping, and TEG6s. Specimens will be transported utilizing Specimen Transport Guidelines.
  Interventions: Other: Laboratory clotting studies

INTERVENTIONS:
Other: Laboratory clotting studies — Cord blood will be utilized to perform lab test including PT, aPTT, fibrinogen, platelet count, platelet mapping, and TEG6s

SUMMARY:
Thromboelastography (TEG) is a laboratory technique used to examine the process of clot formation and degradation by measuring and reporting the kinetic changes, the rate of clot formation, clot strength, and clot stability. TEG provides numeric values and a graphical representation of the primary and secondary hemostatic systems and fibrinolysis more quickly and with a smaller blood sample than routine coagulation studies. TEG6s, the newest TEG platform, simplifies and standardizes TEG technique and is currently available at only four US children's hospitals. Normative values of TEG6s results have not been established in healthy neonates. There are a number of well-established perinatal risk factors for thrombosis in the newborn; however, maternal diabetes has been the most frequently identified risk factor in the newborn since 1965. Despite the well-established hypercoagulable state observed in infants of diabetic mothers (IDMs), there have been no studies evaluating TEG in IDMs. To establish normative data and investigate the hypercoagulable state of IDMs, this observational prospective cohort study will evaluate TEG6s in these two populations: a control group that will include neonates ≥37 weeks gestational age born to mothers with uncomplicated pregnancies and a comparison group that will include neonates ≥37 weeks born to mothers with gestational diabetes or a history of Type 1 or Type 2 diabetes prior to pregnancy, either requiring insulin or diet controlled. We hypothesize that cord blood TEG6s results will differ between healthy newborns and IDMs reflecting a hypercoagulable state in IDMs with an increased coagulation index (CI) in the IDM group. A sample size calculation was performed for a two-sample t-test using the POWER procedure in SAS version 9.4. Based on a two-tailed alpha of 0.05 and a standard deviation of 0.9, the total N was determined to be 40 (i.e., 20 in each group). This yields a power of 0.84 to detect a difference of 1.25 units in the mean CI between IDMs and healthy controls. To avoid blood loss and skin breaking procedures in the subjects, umbilical cord blood obtained from the umbilical cord will be used for analysis. To assure appropriate dilution, a hematocrit will be measured at the time of blood collection using a blood gas machine for prompt results. Sample blood will immediately be taken by the investigators from the delivery hospital to the children's hospital, where the following clotting studies will be performed: PT, aPTT, fibrinogen, platelet count, platelet mapping, and TEG6s. Statistical analyses will be performed on the results of these studies and will provide normative data in healthy newborns and infants of diabetic mothers. Having data on the coagulation profile of neonates will help guide management techniques and help explain the propensity to clot among IDMs and guide further research into prevention and treatment of this complication.

DETAILED DESCRIPTION:
Thromboelastography (TEG), is a laboratory technique used to examine the process of clot formation and degradation by measuring and reporting the kinetic changes, the rate of clot formation, clot strength, and clot stability in umbilical cord blood samples. TEG provides numeric values and a graphical representation of the primary and secondary hemostatic systems and fibrinolysis. The current standard assessments of coagulation status require a combination of multiple tests with multiple blood samples. These tests, including prothrombin time (PT), partial thromboplastin time (aPTT), fibrinogen level, and platelet count, only partially reflect components of the coagulation system, whereas TEG reflects the complex interplay between coagulation factors, cellular components, enzymes, and highly organized feedback mechanisms that maintain equilibrium between clot formation and lysis. TEG has advantages over routine coagulation studies because it is able to assess coagulation function more quickly and with a single smaller blood sample.

A few studies, however, have established normative TEG results in newborns. These studies used older TEG systems/technology. There is a newer TEG6s platform which is currently available at Arkansas Children's Hospital (ACH) and only 3 other children's hospitals in the country. Normative values using TEG6s have not been established in healthy neonates. In fact, although there are investigations in adults, there are no published studies using this newer technology in newborns. The lack of normative standards for TEG6s in newborns is limiting the use of this technology in research and clinical practice.

TEG6s simplifies and standardizes the technique for performing TEG by eliminating the need for manual pipetting. This platform also enables multiple assays to be performed simultaneously from a single blood sample. The TEG6s measures clot viscoelasticity throughout the coagulation process by using resonance technology. Using light-emitting diode illumination, an infrared detector measures vertical motion of the coagulating blood meniscus. Greater clot strength causes higher resonant frequencies, which is subsequently identified by the detector and converted to a graphical image. The TEG6s can deliver the same quality test results without the complicated test preparation process required when using the older TEG platform.

There are a number of well-established perinatal risk factors for thrombosis in the newborn, including systemic infections, dehydration, congenital heart disease, birth asphyxia, polycythemia, presence of intravascular catheters, inherited thrombophilias, and transplacental passage of maternal antiphospholipid and anticardiolipin antibodies. Described since at least 1965, however, maternal diabetes is the most frequently identified risk factor. This risk of thrombosis in infants of diabetic mothers (IDM) has been found to be 15.8% compared with <1% in the non-IDM group. Despite the well-established hypercoagulable state observed in IDMs, there have been no studies evaluating TEG in these newborns.

Currently, there are few published studies on TEG as it relates to neonates. The clotting profile in neonates differs vastly from adults and even the pediatric population, explaining why prior data on TEG from these populations cannot be extrapolated to this special population of newborns. The significant difference is likely explained by the delicate balance in the neonatal hemostatic system that is composed of lower levels of plasma coagulation inhibitors, such as antithrombin, protein C, and protein S, while having procoagulant factor levels, such as factor VIII, von Willebrand factor (vWF), and factor XIII levels that are comparable to the levels in adults.

There have been prior studies establishing normative values for TEG in term newborns but none with the new TEG6s platform. Furthermore, there have been minimal studies looking into the diverse subgroups of the neonatal population on either TEG or TEG6s. With regards to my proposed project, TEG is likely to identify differences among healthy newborns and IDMs, which will help explain the propensity to clot and guide further research into prevention and treatment of this complication.

The study of coagulation currently entails multiple tests, requires multiple blood samples, and has a waiting period for laboratory results. Large volumes of repeated blood sampling in this physically small-sized population can lead to iatrogenic anemia. TEG6s, however, uses a single blood sample to deliver results quickly with both a graphical representation and numeric value. The results provided by TEG are useful in helping to determine specific deficiencies affecting a patient, for example, clotting factors, heparin, fibrinogen and platelets.

ELIGIBILITY:
Inclusion Criteria:

* Control Group: Healthy term neonates

  * Infants born at 37 weeks gestational age or greater born to mothers of any age with uncomplicated pregnancies
* Comparison Group: Term infants of diabetic mothers

  * Infants born at 37 weeks gestational age or greater to mothers of any age with gestational diabetes or Type 1 or Type 2 diabetes, managed with either diet or insulin

Exclusion Criteria:

* For Both Groups:

  * Infants <37 weeks gestational age
  * Multiple gestation pregnancies
  * Maternal thrombocytopenia
  * Known fetal anomalies
  * Known maternal blood clotting disorders or history of thrombosis
  * Known family history of clotting disorders
  * Chorioamnionitis (diagnosed prior to delivery)
* For "Healthy Term Neonates"

  * Intrauterine growth restriction
  * Gestational hypertension, chronic hypertension, pre-eclampsia, and/or eclampsia
  * Any other major complication of pregnancy or major medical history

Ages: 0 Hours to 2 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Mothers delivering or scheduled to deliver at the Labor and Delivery unit at UAMS when study personnel are available will be approached to discuss participation if they meet criteria for enrollment.
  A control group will include neonates ≥37 weeks gestational age on day of life 1 born to mothers with uncomplicated pregnancies and a comparison group that will include neonates ≥37 weeks gestational age on day of life 1 born to mothers with gestational diabetes or a history of Type 1 or Type 2 diabetes prior to pregnancy, either requiring insulin or diet controlled. The control group will include 20 subjects, and the comparison group will include 20 subjects.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2023-01-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Coagulation Index | Data will be obtained at time of delivery on day of life 1
  The coagulation index composed of the various components from TEG6s will be calculated and analyzed by a statistician

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra G Woodle, MD, Principal Investigator — ACHRI
Locations (1):
- Arkansas Children's Hospital, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Edwards RM, Naik-Mathuria BJ, Gay AN, Olutoye OO, Teruya J. Parameters of thromboelastography in healthy newborns. Am J Clin Pathol. 2008 Jul;130(1):99-102. doi: 10.1309/LABNMY41RUD099J2. PMID 18550478
- [Background] Sidlik R, Strauss T, Morag I, Shenkman B, Tamarin I, Lubetsky A, Livnat T, Kenet G. Assessment of Functional Fibrinolysis in Cord Blood Using Modified Thromboelastography. Pediatr Blood Cancer. 2016 May;63(5):839-43. doi: 10.1002/pbc.25865. Epub 2016 Jan 8. PMID 26749087
- [Background] Sewell EK, Forman KR, Wong EC, Gallagher M, Luban NL, Massaro AN. Thromboelastography in term neonates: an alternative approach to evaluating coagulopathy. Arch Dis Child Fetal Neonatal Ed. 2017 Jan;102(1):F79-F84. doi: 10.1136/archdischild-2016-310545. Epub 2016 May 13. PMID 27178714
- [Background] Erdoes G, Schloer H, Eberle B, Nagler M. Next generation viscoelasticity assays in cardiothoracic surgery: Feasibility of the TEG6s system. PLoS One. 2018 Dec 20;13(12):e0209360. doi: 10.1371/journal.pone.0209360. eCollection 2018. PMID 30571781
- [Background] Lloyd-Donald P, Churilov L, Zia F, Bellomo R, Hart G, McCall P, Martensson J, Glassford N, Weinberg L. Assessment of agreement and interchangeability between the TEG5000 and TEG6S thromboelastography haemostasis analysers: a prospective validation study. BMC Anesthesiol. 2019 Mar 30;19(1):45. doi: 10.1186/s12871-019-0717-7. PMID 30927909
- [Background] Sarkar S, Hagstrom NJ, Ingardia CJ, Lerer T, Herson VC. Prothrombotic risk factors in infants of diabetic mothers. J Perinatol. 2005 Feb;25(2):134-8. doi: 10.1038/sj.jp.7211222. PMID 15526010
- [Background] Oppenheimer EH, Esterly JR. Thrombosis in the newborn: comparison between infants of diabetic and nondiabetic mothers. J Pediatr. 1965 Oct;67(4):549-56. doi: 10.1016/s0022-3476(65)80424-3. No abstract available. PMID 5319226